CLINICAL TRIAL: NCT02415335
Title: Dexamethasone Preoperative for Patients Undergoing Laparoscopy for Suspected Appendicitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2014-707; 2014-005040-18 (EudraCT Number)
Record Dates: First submitted 2015-03-31; First posted 2015-04-14 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Suspected Appendicitis
MeSH Terms: interventions — dexamethasone 21-phosphate; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Injection of 2 ml isotonic NaCl intravenously minimum 30 minutes preoperative.
  Interventions: Drug: Isotonic NaCl
- dexamethasone (Experimental): Injection of 2 ml 4 mg/ml dexamethasone phosphate intravenously minimum 30 minutes preoperative.
  Interventions: Drug: dexamethasone phosphate

INTERVENTIONS:
Drug: dexamethasone phosphate — Intravenously administration minimum of 30 minutes preoperatively.
  Other Names: Dexamethasone
  Arms: dexamethasone
Drug: Isotonic NaCl — Intravenously administration minimum of 30 minutes preoperatively
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
For elective abdominal surgery preoperative administration of 8 mg dexamethasone reduces the incidents of postoperative nausea and vomiting (PONV). Whether preoperative administration of 8 mg dexamethasone reduces PONV for patients having acute abdominal surgery has not been established. The investigators wish to see if preoperative administration of 8 mg dexamethasone minimum 30 minutes prior to a diagnostic laparoscopy for suspected appendicitis will reduce the incidents of PONV by 50%. Of secondary interest the investigators want to see if 8 mg dexamethasone preoperative can reduce pain, reduce opioid consumption, postoperative fatigue, duration of time until resumption of work and resumption of normal daily activities, and enhanced the quality of recovery.

DETAILED DESCRIPTION:
Eligible patients undergoing a diagnostic laparoscopy for suspected appendicitis will be randomized to receive placebo or 8 mg dexamethasone intravenously minimum 30 minutes prior to the operation.

Randomization will be done by envelope randomization. We would expect that 60% of the patients would experience postoperative nausea or vomiting (PONV) during the first 24-32 hours postoperatively. To show a 50% reduction in the incidents of PONV during the first 24-32 hours postoperatively (with a power of 80%, a significant level of 5% and a loss to follow up of 20%) we need 60 patients in each arm. So a total of 120 patients are to be randomized 1:1.

Both sites use paper Case Report Forms (CRF). The trial will be monitored by the regional GCP (Good Clinical Practice) unit and adhere to GCP guidelines.

Patients are assessed by self reporting questionnaires preoperatively and postoperatively after 2-10 hours, 8-16 hours, 24-32 hours, on postoperative day (POD) 2, POD 3, POD 7, POD 14 and POD 30.

Preoperative anxiety recorded by a VAS scale, Pain Catastrophizing Scale and Hospital anxiety and depression scale are recorded by the preoperative questionnaire.

A short telephone interview will be done during the first postoperative day regarding duration of abdominal pain prior to admission, social status regarding children and whether they living with another adult, smoking status, use of sleep medication or use of psychopharmacy a minimum of 7 days prior to the operation, physical level of normal daily activities, physical level of work, educational and occupational background.

Other demographics such as height, weight, ASA class, age, last CRP prior to the operation, duration of the operation, date and time of admission, date and time of discharge are registered through the electronic patient record files. Pathology of any removed tissue are registered trough the pathology report.

Diagnosis at the operation, preformed procedure, whether the preforming surgeon was supervised, number of identical procedures preformed previous by the surgeon or the surgeons supervisor (if supervised) will be recorded in the patients CRF by the preforming surgeon.

Pre-, intra- and post-operative pain medication, antiemetics and antibiotics are recorded through the electronic patient medication files.

Postoperative complications and adverse events are recorded through the electronic patient record files and by telephone interview.

To ensure a high completion rate, patients are contacted by telephone at each registration time postoperatively.

Parametric or non-parametric statistical analysis will be used when appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for a diagnostic laparoscopy for suspected appendicitis
* ASA clas I-III

Exclusion Criteria:

* Known inflammatory bowel disease
* Known autoimmune disease.
* Chronic pain patient.
* Pregnant or breastfeeding.
* In treatment with systemic corticoid steroids or immune-depressants.
* Known glaucoma.
* Known ocular herpes simplex.
* Vaccination within 14 days prior to inclusion.
* Known cushing's disease.
* Known myasthenia gravis.
* Presumably poor compliance with study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2015-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting (PONV) | 24-32 hours postoperative
  Incidents of nausea and/or vomiting during the first 24-32 hours postoperative

SECONDARY OUTCOMES:
Pain at rest (VAS scale) | 2-10 hours postoperative
  Pain at rest measured on a 100 mm VAS scale
Pain when coughing (VAS scale) | 2-10 hours postoperative
  Pain when coughing measured on a 100 mm VAS scale
Postoperative fatigue (VAS scale) | 2-10 hours postoperative
  Postoperative fatigue measured on a 100 mm VAS scale
Quality of recovery (QoR-15D questionnaire) | 24-32 hours postoperative
  Quality of recovery measured by the QoR-15D questionnaire
Time until resumption of normal daily activities | Registration when resumption, expected to be within 60 days postoperatively
  Time until resumption of normal daily activities and reason for not resuming activities earlier
Time until resumption of work | Registration when resumption, expected to be within 60 days postoperatively
  Time until resumption of work and reason for not resuming work earlier
Sleep quality (VAS scale) | 24-32 hours postoperative
  Quality of sleep measured on a 100 mm VAS scale
Postoperative complications (Clavien-Dindo classification of surgical complications) | 30 days postoperative
  30 days postoperative complication according to the Clavien-Dindo classification of surgical complications
Duration of admission | 30 days
  Duration of primary admission
PONV | 2-10 hours postoperatively
PONV | 8-16 hours postoperatively
PONV | 24-32 hours postoperatively
Pain at rest (VAS scale) | 8-16 hours postoperative
  Pain at rest measured on a 100 mm VAS scale
Pain at rest (VAS scale) | 24-32 hours postoperative
  Pain at rest measured on a 100 mm VAS scale
Pain at rest (VAS scale) | POD (Post Operative Day) 2
  Pain at rest measured on a 100 mm VAS scale
Pain at rest (VAS scale) | POD3
  Pain at rest measured on a 100 mm VAS scale
Pain at rest (VAS scale) | POD7
  Pain at rest measured on a 100 mm VAS scale
Pain at rest (VAS scale) | POD14
  Pain at rest measured on a 100 mm VAS scale
Pain at rest (VAS scale) | POD30
  Pain at rest measured on a 100 mm VAS scale
Pain when coughing (VAS scale) | 8-16 hours postoperative
  Pain when coughing measured on a 100 mm VAS scale
Pain when coughing (VAS scale) | 24-42 hours postoperative
  Pain when coughing measured on a 100 mm VAS scale
Pain when coughing (VAS scale) | POD2
  Pain when coughing measured on a 100 mm VAS scale
Pain when coughing (VAS scale) | POD3
  Pain when coughing measured on a 100 mm VAS scale
Pain when coughing (VAS scale) | POD7
  Pain when coughing measured on a 100 mm VAS scale
Pain when coughing (VAS scale) | POD14
  Pain when coughing measured on a 100 mm VAS scale
Pain when coughing (VAS scale) | POD30
  Pain when coughing measured on a 100 mm VAS scale
Postoperative fatigue (VAS scale) | 8-16 hours postoperative
  Postoperative fatigue measured on a 100 mm VAS scale
Postoperative fatigue (VAS scale | 24-32 hours postoperative
  Postoperative fatigue measured on a 100 mm VAS scale
Postoperative fatigue (VAS scale | POD2
  Postoperative fatigue measured on a 100 mm VAS scale
Postoperative fatigue (VAS scale | POD3
  Postoperative fatigue measured on a 100 mm VAS scale
Postoperative fatigue (VAS scale | POD7
  Postoperative fatigue measured on a 100 mm VAS scale
Postoperative fatigue (VAS scale | POD14
  Postoperative fatigue measured on a 100 mm VAS scale
Postoperative fatigue (VAS scale | POD30
  Postoperative fatigue measured on a 100 mm VAS scale
Quality of recovery (QoR-15D questionnaire) | POD2
  Quality of recovery measured by the QoR-15D questionnaire
Quality of recovery (QoR-15D questionnaire) | POD3
  Quality of recovery measured by the QoR-15D questionnaire
Quality of recovery (QoR-15D questionnaire) | POD7
  Quality of recovery measured by the QoR-15D questionnaire
Quality of recovery (QoR-15D questionnaire) | POD14
  Quality of recovery measured by the QoR-15D questionnaire
Quality of recovery (QoR-15D questionnaire) | POD30
  Quality of recovery measured by the QoR-15D questionnaire
Sleep quality (VAS scale) | POD2
  Quality of sleep measured on a 100 mm VAS scale
Sleep quality (VAS scale) | POD3
  Quality of sleep measured on a 100 mm VAS scale
Sleep quality (VAS scale) | POD7
  Quality of sleep measured on a 100 mm VAS scale
Sleep quality (VAS scale) | POD14
  Quality of sleep measured on a 100 mm VAS scale
Sleep quality (VAS scale) | POD30
  Quality of sleep measured on a 100 mm VAS scale

OTHER OUTCOMES:
Mobilisation postoperative (Ability to get out of bed) | 2-10 hours postoperative
  Ability to get out of bed
Pain localization (Localization of postoperative pain) | 2-10 hours postoperative
  Localization of postoperative pain
Adverse events | 30 days
  AE, AR, SAR and SUSARS
Mobilisation postoperative (Ability to get out of bed) | 8-16 hours postoperative
  Ability to get out of bed
Mobilisation postoperative (Ability to get out of bed) | 24-32 hours postoperative
  Ability to get out of bed
Pain localization (Localization of postoperative pain) | 8-16 hours postoperative
  Localization of postoperative pain
Pain localization (Localization of postoperative pain) | 24-32 hours postoperative
  Localization of postoperative pain
Pain localization (Localization of postoperative pain) | POD2
  Localization of postoperative pain
Pain localization (Localization of postoperative pain) | POD3
  Localization of postoperative pain
Pain localization (Localization of postoperative pain) | POD7
  Localization of postoperative pain
Pain localization (Localization of postoperative pain) | POD14
  Localization of postoperative pain
Pain localization (Localization of postoperative pain) | POD30
  Localization of postoperative pain

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Kleif, M.D., Principal Investigator — Nordsjaellands Hospital
Locations (2):
- Denmark (2):
  - Kirurgisk afdeling, Nordsjællands Hospital, Hillerød
  - Kirurgisk afdeling, Køge sygehus, Køge

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kleif J, Gogenur I. Severity classification of the quality of recovery-15 score-An observational study. J Surg Res. 2018 May;225:101-107. doi: 10.1016/j.jss.2017.12.040. Epub 2018 Feb 21. PMID 29605019
- [Derived] Kleif J, Kirkegaard A, Vilandt J, Gogenur I. Randomized clinical trial of preoperative dexamethasone on postoperative nausea and vomiting after laparoscopy for suspected appendicitis. Br J Surg. 2017 Mar;104(4):384-392. doi: 10.1002/bjs.10418. Epub 2017 Jan 10. PMID 28072446